CLINICAL TRIAL: NCT03220217
Title: A Multicentre, Randomised, Dose-confirmation, Factorial Phase II Study to Evaluate the Optimal Dose of 68Ga-OPS202 as a PET Imaging Agent in Subjects With Gastroenteropancreatic Neuroendocrine Tumour (GEP-NET)
Brief Title: To Evaluate the Optimal Dose of 68Ga-OPS202 as a PET (Positron Emission Tomography) Imaging Agent in Subjects With Gastroenteropancreatic Neuroendocrine Tumour (GEP-NET)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Diagnostic
Other Study IDs: D-FR-01070-002; 2016-004928-39 (EudraCT Number)
Record Dates: First submitted 2017-06-26; First posted 2017-07-18 (Actual); Results first posted 2021-01-14 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Gastro-Enteropancreatic Neuroendocrine Tumor
MeSH Terms: conditions — Gastro-enteropancreatic neuroendocrine tumor

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: All the primary and secondary imaging endpoints are read by third-party independent readers. Most of the reading will be conducted in blinded manner.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 5-20μg/40-80 MBq, 30-45μg/100-140 MBq (Experimental): Subjects will receive a first intravenous (i.v.) injection of satoreotide trizoxetan with a peptide mass dose range of 5 to 20 μg and a radioactivity dose range 40 to 80 MBq. After 15 to 21 days the subjects will receive a second i.v. injection of satoreotide trizoxetan with a peptide mass dose range of 30-45 μg and a radioactivity dose range 100 to 140 MBq.
  Interventions: Drug: Satoreotide trizoxetan 5-20μg; Drug: Satoreotide trizoxetan 30-45μg
- 5-20μg/100-140 MBq, 30-45μg/160-200 MBq (Experimental): Subjects will receive a first i.v. injection of satoreotide trizoxetan with a peptide mass dose range of 5 to 20 μg and a radioactivity dose range 100 to 140 MBq. After 15 to 21 days the subjects will receive a second i.v. injection of satoreotide trizoxetan with a peptide mass dose range of 30-45 μg and a radioactivity dose range 160 to 200 MBq.
  Interventions: Drug: Satoreotide trizoxetan 5-20μg; Drug: Satoreotide trizoxetan 30-45μg
- 5-20μg/160-200 MBq, 30-45μg/40-80 MBq (Experimental): Subjects will receive a first i.v. injection of satoreotide trizoxetan with a peptide mass dose range of 5 to 20 μg and a radioactivity dose range 160 to 200 MBq. After 15 to 21 days the subjects will receive a second i.v. injection of satoreotide trizoxetan with a peptide mass dose range of 30-45 μg and a radioactivity dose range 40 to 80 MBq.
  Interventions: Drug: Satoreotide trizoxetan 5-20μg; Drug: Satoreotide trizoxetan 30-45μg

INTERVENTIONS:
Drug: Satoreotide trizoxetan 5-20μg — Positron emission tomography (PET) imaging agent
  Other Names: 68Ga-OPS202 5-20μg, 68Ga-IPN01070 5-20μg
Drug: Satoreotide trizoxetan 30-45μg — Positron emission tomography (PET) imaging agent
  Other Names: 68Ga-OPS202 30-45μg, 68Ga-IPN01070 30-45μg

SUMMARY:
The purpose of this clinical research is to confirm the optimal dose of 68Ga-satoreotide trizoxetan (68Ga-IPN01070), formerly 68Ga-OPS202, as a PET imaging agent to be used to detect and localize gastro-entero-pancreatic neuroendocrine tumors (GEP-NETs). 68Ga-IPN01070 is a radiolabelled imaging agent to be used in association with Positron-Emission-Tomography (PET). 68Ga-IPN01070 is made of two main components: 1) IPN01070, an antagonistic somatostatin analogue which binds to the somatostatin receptor (type 2) present on the surface of the tumor cells and 2) Gallium-68, a radioisotope that combined with IPN01070 can be seen in the PET scanner.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed, well differentiated functioning or non-functioning metastatic GEP-NET (Grade I and II as per World Health Organisation classification 2010)
* Confirmed presence of somatostatin receptors (type 2) on technically evaluable tumour lesions documented by a positive Somatostatin Receptor Scan acquired within 6 months prior to screening (Visit 1) and showing minimally two lesions in at least one of the key organs; these images shall be available to be sent to the imaging core lab electronically to ascertain quality and admissibility
* Body weight between 50 kg (110 lb) and 110 kg (243 lb), inclusive
* Adequate bone marrow, liver and renal function
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2

Exclusion Criteria:

* Fewer than five lesions in total and more than 25 lesions/organ detected by the previous somatostatin receptor scan in key organs: liver, lymph nodes, bone or lungs
* Subject who have received treatment of any somatostatin analogue, including Somatuline® Autogel® /Depot®, Sandostatin® LAR within 28 days, and Sandostatin® within 24 hours prior to first 68Ga-OPS202 administration
* Prior or planned administration of a radiopharmaceutical within 8 half-lives of the radionuclide
* Any condition that precludes the proper performance of PET and/or CT scan: a) Subjects who are not able to tolerate the CT contrast agent, b) Subjects with metal implants or arthroplasty, or any other objects that might interfere with the PET and/or CT analysis, c) Subjects unable to raise arms for prolonged imaging purposes, d) Subjects unable to lie still for the entire imaging time, e) Subjects weighing greater than 110 kg (243 lb)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2017-09-26 (Actual); Primary Completion 2019-07-25 (Actual); Study Completion 2019-08-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (5):
- UCLA Medical Center, Los Angeles, California, United States
- Austria (2):
  - Medical University of Innsbruck, Innsbruck
  - University Clinic for Radiology and Nuclear Medicine, Vienna
- Denmark (2):
  - Aarhus University Hospital, Aarhus
  - Rigshospitalet, University of Copenhagen, Copenhagen

REFERENCES:
- [Derived] Miller CG, Gronbaek H, Virgolini I, Kjaer A, Terve P, Bahri S, Iversen P, Svirydenka H, Rohban T, McEwan S. A novel read methodology to evaluate the optimal dose of 68Ga-satoreotide trizoxetan as a PET imaging agent in patients with gastroenteropancreatic neuroendocrine tumours: a phase II clinical trial. EJNMMI Res. 2021 Sep 6;11(1):84. doi: 10.1186/s13550-021-00819-1. PMID 34487283

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This dose-confirmation study was conducted at 4 centres between September 2017 and August 2019. Adult subjects with somatostatin receptor subtype 2 (sstr2)-positive gastroenteropancreatic neuroendocrine tumour (GEP-NET) were randomised to investigational imaging product with Gallium-68 (68Ga)-satoreotide trizoxetan (68Ga-IPN01070, formerly known as 68Ga-OPS202).
Pre-assignment Details: The Screening Visit (Visit 1) was performed within 2 weeks prior to the first 68Ga-satoreotide trizoxetan administration. Subjects' eligibility was re-checked by the investigator at Visit 2 (Day 1) before randomisation to 1 of 3 study arms (A, B or C) with differing 68Ga-satoreotide trizoxetan peptide mass dose and radioactivity dose range combinations.
Groups:
- Arm A: 5-20 µg/40-80 MBq Then 30-45 µg/100-140 MBq: Subjects received a single intravenous (i.v.) injection of 68Ga-satoreotide trizoxetan with a peptide mass dose range of 5-20 micrograms (μg) and a radioactivity dose range of 40-80 Megabecquerel (MBq) on Visit 2 (Day 1).
  After 15 to 21 days at Visit 3 (Days 16 to 22), subjects received a second i.v. injection of 68Ga-satoreotide trizoxetan with a peptide mass dose range of 30-45 μg and a radioactivity dose range of 100-140 MBq.
  Both injections were followed by positron emission tomography(PET)/computed tomography (CT) scan imaging 1 hour post dosing (up to 80 min).
- Arm B: 5-20 µg/100-140 MBq Then 30-45 µg/160-200 MBq: Subjects received a single i.v. injection of 68Ga-satoreotide trizoxetan with a peptide mass dose range of 5-20 μg and a radioactivity dose range of 100-140 MBq on Visit 2 (Day 1).
  After 15 to 21 days at Visit 3 (Days 16 to 22), subjects received a second i.v. injection of 68Ga-satoreotide trizoxetan with a peptide mass dose range of 30-45 μg and a radioactivity dose range of 160-200 MBq.
  Both injections were followed by PET/CT scan imaging 1 hour post dosing (up to 80 min).
- Arm C: 5-20 µg/160-200 MBq Then 30-45 µg/40-80 MBq: Subjects received a single i.v. injection of 68Ga-satoreotide trizoxetan with a peptide mass dose range of 5-20 μg and a radioactivity dose range of 160-200 MBq on Visit 2 (Day 1).
  After 15 to 21 days at Visit 3 (Days 16 to 22), subjects received a second i.v. injection of 68Ga-satoreotide trizoxetan with a peptide mass of 30-45 μg and a radioactivity range of 40-80 MBq.
  Both injections were followed by PET/CT scan imaging 1 hour post dosing (up to 80 min).
Period: Overall Study
Arm/Group | Arm A: 5-20 µg/40-80 MBq Then 30-45 µg/100-140 MBq | Arm B: 5-20 µg/100-140 MBq Then 30-45 µg/160-200 MBq | Arm C: 5-20 µg/160-200 MBq Then 30-45 µg/40-80 MBq
Started (Received 68Ga-satoreotide trizoxetan) | 8 | 10 | 11
Completed (Completed Study) | 8 | 9 | 10
Not Completed | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Subject Missed Procedure | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The randomised population included all subjects randomly assigned to a dosing arm/sequence.
Groups:
- Arm A: 5-20 µg/40-80 MBq Then 30-45 µg/100-140 MBq: Subjects received a single i.v. injection of 68Ga-satoreotide trizoxetan with a peptide mass dose range of 5-20 μg and a radioactivity dose range of 40-80 MBq on Visit 2 (Day 1).
  After 15 to 21 days at Visit 3 (Days 16 to 22), subjects received a second i.v. injection of 68Ga-satoreotide trizoxetan with a peptide mass dose range of 30-45 μg and a radioactivity dose range of 100-140 MBq.
  Both injections were followed by PET/CT scan imaging 1 hour post dosing (up to 80 min).
- Arm C: 5-20 µg/160-200 MBq Then 30-45 µg/40-80 MBq: Subjects received a single i.v. injection of 68Ga-satoreotide trizoxetan with a peptide mass dose range of 5-20 μg and a radioactivity dose range of 160-200 MBq on Visit 2 (Day 1).
  After 15 to 21 days at Visit 3 (Days 16 to 22), subjects received a second i.v. injection of 68Ga-satoreotide trizoxetan with a peptide mass dose range of 30-45 μg and a radioactivity range of 40-80 MBq.
  Both injections were followed by PET/CT scan imaging 1 hour post dosing (up to 80 min).
- Total: Total of all reporting groups
Arm/Group | Arm A: 5-20 µg/40-80 MBq Then 30-45 µg/100-140 MBq | Arm B: 5-20 µg/100-140 MBq Then 30-45 µg/160-200 MBq | Arm C: 5-20 µg/160-200 MBq Then 30-45 µg/40-80 MBq | Total
Number analyzed (Participants) | 8 | 10 | 11 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 4 | 8 | 15
  >=65 years | 5 | 6 | 3 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.5 (11.1) | 67.6 (6.4) | 60.7 (12.3) | 65.8 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 6 | 2 | 10
  Male | 6 | 4 | 9 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1
  White | 8 | 10 | 10 | 28
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Relative Lesion Counts Presented by Combination of Injected Peptide/Radioactivity Dose Ranges
Description: For each combination of injected peptide/radioactivity dose range, relative lesion counts were measured as the ratio of the number of lesions detected by 68Ga-satoreotide trizoxetan PET/CT and PET readings to the number of lesions assessed by standard-of-truth (SoT). The SoT in this study was the contrast enhanced (ce)CT scan images acquired at Visit 2 (Day 1) and Visit 3 (Days 16 to 22). Relative lesion counts for PET/CT and PET readings are presented for all organs, primary site of GEP-NET and per organ by each combination of injected peptide/radioactivity dose range after the 1st and 2nd injections.
Time Frame: Day 1 and Days 16 to 22
Population: Results are presented for the Per Protocol (PP) population which consisted of the first 24 randomised subjects who could be assessed and for whom no major protocol violations/deviations impacting primary endpoint results occurred. Only subjects with data available were included in the analysis.
Measure: Median (Full Range); unit: Ratio
Groups:
- Arm A: 5-20 μg/40-80 MBq: Subjects received a single i.v. injection of 68Ga-satoreotide trizoxetan with a peptide mass of 5-20 μg and a radioactivity range of 40-80 MBq on Visit 2/Day 1.
- Arm A: 30-45 μg/100-140 MBq: Subjects received a single i.v. injection of 68Ga-satoreotide trizoxetan with a peptide mass of 30-45 μg and a radioactivity range of 100-140 MBq on Visit 3/Days 16 to 22.
- Arm B: 5-20 μg/100-140 MBq: Subjects received a single i.v. injection of 68Ga-satoreotide trizoxetan with a peptide mass of 5-20 μg and a radioactivity range of 100-140 MBq on Visit 2/Day 1.
- Arm B: 30-45 μg/160-200 MBq: Subjects received a single i.v. injection of 68Ga-satoreotide trizoxetan with a peptide mass of 30-45 μg and a radioactivity range of 160-200 MBq on Visit 3/Days 16 to 22.
- Arm C: 5-20 μg/160-200 MBq: Subjects received a single i.v. injection of 68Ga-satoreotide trizoxetan with a peptide mass of 5-20 μg and a radioactivity range of 160-200 MBq on Visit 2/Day 1.
- Arm C: 30-45 μg/40-80 MBq: Subjects received a single i.v. injection of 68Ga-satoreotide trizoxetan with a peptide mass of 30-45 μg and a radioactivity range of 40-80 MBq on Visit 3/Days 16 to 22.
Arm/Group | Arm A: 5-20 μg/40-80 MBq | Arm A: 30-45 μg/100-140 MBq | Arm B: 5-20 μg/100-140 MBq | Arm B: 30-45 μg/160-200 MBq | Arm C: 5-20 μg/160-200 MBq | Arm C: 30-45 μg/40-80 MBq
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8
Ratio
  PET/CT: All Organs | 3.6 [0.73 to 15.00] | 3.8 [1.71 to 13.50] | 2.1 [0.64 to 4.41] | 2.6 [0.82 to 5.25] | 2.7 [0.91 to 16.25] | 2.5 [0.82 to 9.75]
  PET/CT: Primary Site: number analyzed (Participants) | 2 | 2 | 2 | 2 | 1 | 1
  PET/CT: Primary Site | 0.8 [0.50 to 1.00] | 0.8 [0.50 to 1.00] | 0.5 [0.00 to 1.00] | 1.0 [1.00 to 1.00] | 1.0 [1.00 to 1.00] | 1.0 [1.00 to 1.00]
  PET/CT: Liver: number analyzed (Participants) | 5 | 5 | 4 | 4 | 8 | 8
  PET/CT: Liver | 2.1 [0.73 to 9.00] | 3.0 [2.00 to 8.00] | 2.9 [0.83 to 8.00] | 3.5 [1.50 to 11.00] | 2.4 [0.86 to 7.5] | 2.6 [0.76 to 5.17]
  PET/CT: Lymph Nodes: number analyzed (Participants) | 3 | 3 | 6 | 6 | 4 | 4
  PET/CT: Lymph Nodes | 2.0 [1.80 to 3.00] | 2.0 [0.40 to 3.00] | 1.00 [0.00 to 8.00] | 0.9 [0.00 to 12.00] | 2.2 [1.25 to 5.00] | 1.6 [1.00 to 2.00]
  PET/CT: Bone: number analyzed (Participants) | 0 | 0 | 1 | 1 | 0 | 0
  PET/CT: Bone |  |  | 4.6 [4.6 to 4.6] | 3.6 [3.6 to 3.6] |  |
  PET/CT: Lung: number analyzed (Participants) | 0 | 0 | 2 | 2 | 0 | 0
  PET/CT: Lung |  |  | 0.5 [0.00 to 1.00] | 1.0 [0.00 to 2.00] |  |
  PET: All Organs | 2.6 [0.73 to 19.00] | 3.9 [1.00 to 14.50] | 2.2 [1.00 to 4.50] | 2.6 [1.50 to 4.75] | 2.8 [0.91 to 13.50] | 2.7 [0.68 to 7.50]
  PET: Primary Site: number analyzed (Participants) | 2 | 2 | 2 | 2 | 1 | 1
  PET: Primary Site | 0.8 [0.50 to 1.00] | 0.8 [0.50 to 1.00] | 1.0 [1.00 to 1.00] | 0.5 [0.00 to 1.00] | 1.0 [1.00 to 1.00] | 1.0 [1.00 to 1.00]
  PET: Liver: number analyzed (Participants) | 5 | 5 | 4 | 4 | 8 | 8
  PET: Liver | 2.6 [0.73 to 5.00] | 3.3 [1.00 to 7.00] | 2.9 [0.67 to 7.00] | 3.4 [1.33 to 9.00] | 2.4 [0.86 to 7.00] | 2.3 [0.62 to 6.00]
  PET: Lymph Nodes: number analyzed (Participants) | 3 | 3 | 6 | 3 | 4 | 4
  PET: Lymph Nodes | 2.0 [1.80 to 3.00] | 2.0 [1.60 to 4.00] | 2.2 [0.50 to 10.0] | 2.0 [0.50 to 14.00] | 3.8 [1.00 to 6.00] | 3.1 [0.75 to 4.00]
  PET: Bone: number analyzed (Participants) | 0 | 0 | 1 | 1 | 0 | 0
  PET: Bone |  |  | 3.6 [3.6 to 3.6] | 3.8 [3.8 to 3.8] |  |
  PET: Lung: number analyzed (Participants) | 0 | 0 | 2 | 2 | 0 | 0
  PET: Lung |  |  | 0.5 [0.00 to 1.00] | 1.5 [0.00 to 3.00] |  |

2. Primary Outcome: Relative Lesion Counts Presented by Peptide Mass and Radioactivity Dose Ranges
Description: For each combination of injected peptide/radioactivity dose range, relative lesion counts were measured as the ratio of the number of lesions detected by 68Ga-satoreotide trizoxetan PET/CT and PET readings to the number of lesions assessed by SoT. The SoT in this study was the ceCT scan images acquired at Visit 2 (Day 1) and Visit 3 (Day 16 to 22). Relative lesion counts for PET/CT and PET readings are presented for all organs, primary site of GEP-NET and per organ by both peptide mass range and radioactivity dose range.
Time Frame: Day 1 and Days 16 to 22
Population: Results are presented for the PP population which consisted of the first 24 randomised subjects who could be assessed and for whom no major protocol violations/deviations impacting primary endpoint results occurred. Only subjects with data available were included in the analysis.
Measure: Median (Full Range); unit: Ratio
Groups:
- Peptide Mass Dose Range 5-20 μg: Subjects from Arms A, B and C who received an injection of 68Ga-satoreotide trizoxetan with a peptide mass dose range of 5-20 μg on Visit 2 (Day 1).
- Peptide Mass Dose Range 30-45 μg: Subjects from Arms A, B and C who received an injection of 68Ga-satoreotide trizoxetan with a peptide mass dose range of 30-45 μg on Visit 3 (Days 16-22).
- Radioactivity Dose Range 40-80 MBq: Subjects from Arms A and C who received an injection of 68Ga-satoreotide trizoxetan with a radioactivity dose of 40-80 MBq on either Visit 2 (Day 1) or on Visit 3 (Days 16-22).
- Radioactivity Dose Range 100-140 MBq: Subjects from Arms A and B who received an injection of 68Ga-satoreotide trizoxetan with a radioactivity dose range of 100-140 MBq on either Visit 2(Day 1) or on Visit 3 (Days 16-22).
- Radioactivity Dose Range 160-200 MBq: Subjects from Arms B and C who received an injection of 68Ga-satoreotide trizoxetan with a radioactivity dose range of 160-200 MBq on either Visit 2 (Day 1) or on Visit 3 (Days 16-22).
Arm/Group | Peptide Mass Dose Range 5-20 μg | Peptide Mass Dose Range 30-45 μg | Radioactivity Dose Range 40-80 MBq | Radioactivity Dose Range 100-140 MBq | Radioactivity Dose Range 160-200 MBq
Number analyzed (Participants) | 24 | 24 | 16 | 16 | 16
Ratio
  PET/CT: All Organs | 2.7 [0.64 to 16.25] | 2.7 [0.82 to 13.50] | 3.1 [0.73 to 15.00] | 2.6 [0.64 to 13.50] | 2.6 [0.82 to 16.25]
  PET/CT: Primary Site: number analyzed (Participants) | 5 | 5 | 3 | 4 | 3
  PET/CT: Primary Site | 1.0 [0.00 to 1.00] | 1.0 [0.50 to 1.00] | 1.0 [0.50 to 1.00] | 0.8 [0.00 to 1.00] | 1.0 [1.00 to 1.00]
  PET/CT: Liver: number analyzed (Participants) | 17 | 17 | 13 | 9 | 12
  PET/CT: Liver | 2.3 [0.73 to 9.00] | 3.0 [0.76 to 11.00] | 2.2 [0.73 to 9.00] | 3.0 [0.83 to 8.00] | 2.7 [0.86 to 11.00]
  PET/CT: Lymph Nodes: number analyzed (Participants) | 13 | 13 | 7 | 9 | 10
  PET/CT: Lymph Nodes | 2.0 [0.00 to 8.00] | 1.3 [0.00 to 12.00] | 2.0 [1.00 to 3.00] | 1.3 [0.00 to 8.00] | 1.3 [0.00 to 12.00]
  PET/CT: Bone: number analyzed (Participants) | 1 | 1 | 0 | 1 | 1
  PET/CT: Bone | 4.6 [4.6 to 4.6] | 3.6 [3.6 to 3.6] |  | 4.6 [4.6 to 4.6] | 3.6 [3.6 to 3.6]
  PET/CT: Lung: number analyzed (Participants) | 2 | 2 | 0 | 2 | 2
  PET/CT: Lung | 0.5 [0.00 to 1.00] | 1.0 [0.00 to 2.00] |  | 0.5 [0.00 to 1.00] | 1.0 [0.00 to 2.00]
  PET: All Organs | 2.6 [0.73 to 19.00] | 2.8 [0.68 to 14.50] | 2.6 [0.68 to 19.00] | 2.8 [1.00 to 14.50] | 2.7 [0.91 to 13.50]
  PET: Primary Site: number analyzed (Participants) | 5 | 5 | 3 | 4 | 3
  PET: Primary Site | 1.0 [0.50 to 1.00] | 1.0 [0.00 to 1.00] | 1.0 [0.50 to 1.00] | 1.0 [0.50 to 1.00] | 1.0 [0.00 to 1.00]
  PET: Liver: number analyzed (Participants) | 17 | 17 | 13 | 9 | 12
  PET: Liver | 2.6 [0.67 to 7.00] | 2.8 [0.62 to 9.00] | 2.6 [0.62 to 6.00] | 3.3 [0.67 to 7.00] | 2.8 [0.86 to 9.00]
  PET: Lymph Nodes: number analyzed (Participants) | 13 | 13 | 7 | 9 | 10
  PET: Lymph Nodes | 2.3 [0.50 to 10.00] | 2.0 [0.50 to 14.00] | 2.7 [0.75 to 4.00] | 2.0 [0.50 to 10.00] | 2.2 [0.50 to 14.00]
  PET: Bone: number analyzed (Participants) | 1 | 1 | 0 | 1 | 1
  PET: Bone | 3.6 [3.6 to 3.6] | 3.8 [3.8 to 3.8] |  | 3.6 [3.6 to 3.6] | 3.8 [3.8 to 3.8]
  PET: Lung: number analyzed (Participants) | 2 | 2 | 0 | 2 | 2
  PET: Lung | 0.5 [0.00 to 1.00] | 1.5 [0.00 to 3.00] |  | 0.5 [0.00 to 1.00] | 1.5 [0.00 to 3.00]

3. Secondary Outcome: Image Quality as Assessed by Tumour-To-Background Ratio Presented by Combination of Injected Peptide/Radioactivity Dose Range
Description: For each PET assessment, image quality was quantitatively measured by the tumour-to-background ratio, obtained using the mean of all lesions tumour-to-backgrounds, for each of the following organs; liver, lymph nodes, bone and lungs. The tumour-to-background ratio was computed by mean standardised uptake value (SUVmean) of the lesion divided by the SUVmean of the subject's reference tissue (tumour-free liver or aortic blood). A high tumour-to-background ratio indicates high effectiveness of 68Ga-satoreotide trizoxetan as a diagnostic agent. Tumour-to-background ratios are presented for primary site of GEP-NET and per organ by each combination of injected peptide/radioactivity dose range.
Time Frame: Day 1 and Days 16 to 22
Population: as for outcome 2
Measure: Median (Full Range); unit: Ratio
Groups:
- Arm A: 5-20 μg/40-80 MBq: Subjects received a single i.v. injection of 68Ga-satoreotide trizoxetan with a peptide mass dose range of 5-20 μg and a radioactivity range of 40-80 MBq on Visit 2 (Day 1).
- Arm A: 30-45 μg/100-140 MBq: Subjects received a single i.v. injection of 68Ga-satoreotide trizoxetan with a peptide mass dose range of 30-45 μg and a radioactivity range of 100-140 MBq on Visit 3 (Days 16 to 22).
- Arm B: 5-20 μg/100-140 MBq: Subjects received a single i.v. injection of 68Ga-satoreotide trizoxetan with a peptide mass dose range of 5-20 μg and a radioactivity range of 100-140 MBq on Visit 2 (Day 1).
- Arm B: 30-45 μg/160-200 MBq: Subjects received a single i.v. injection of 68Ga-satoreotide trizoxetan with a peptide mass dose range of 30-45 μg and a radioactivity range of 160-200 MBq on Visit 3 (Days 16 to 22).
- Arm C: 5-20 μg/160-200 MBq: Subjects received a single i.v. injection of 68Ga-satoreotide trizoxetan with a peptide mass dose range of 5-20 μg and a radioactivity range of 160-200 MBq.
- Arm C: 30-45 μg/40-80 MBq: Subjects received a single i.v. injection of 68Ga-satoreotide trizoxetan with a peptide mass dose range of 30-45 μg and a radioactivity range of 40-80 MBq on Visit 3 (Days 16 to 22).
Arm/Group | Arm A: 5-20 μg/40-80 MBq | Arm A: 30-45 μg/100-140 MBq | Arm B: 5-20 μg/100-140 MBq | Arm B: 30-45 μg/160-200 MBq | Arm C: 5-20 μg/160-200 MBq | Arm C: 30-45 μg/40-80 MBq
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8
Ratio
  Primary Site: number analyzed (Participants) | 2 | 2 | 3 | 2 | 1 | 1
  Primary Site | 26.4 [7.04 to 45.84] | 17.5 [7.07 to 27.87] | 4.8 [4.57 to 33.81] | 18.1 [3.29 to 32.81] | 2.3 [2.3 to 2.3] | 2.2 [2.2 to 2.2]
  Liver: number analyzed (Participants) | 5 | 5 | 5 | 5 | 8 | 8
  Liver | 5.5 [3.75 to 12.88] | 4.7 [3.56 to 9.96] | 4.2 [3.10 to 24.95] | 4.2 [3.05 to 29.33] | 3.6 [2.13 to 10.75] | 4.0 [3.07 to 22.48]
  Lymph Nodes: number analyzed (Participants) | 3 | 3 | 6 | 6 | 5 | 5
  Lymph Nodes | 7.4 [3.87 to 16.98] | 6.2 [3.22 to 13.76] | 5.1 [2.55 to 16.10] | 8.2 [1.54 to 13.70] | 5.7 [3.40 to 12.84] | 4.5 [3.50 to 18.69]
  Bone: number analyzed (Participants) | 0 | 0 | 1 | 1 | 0 | 0
  Bone |  |  | 12.7 [12.7 to 12.7] | 9.2 [9.2 to 9.2] |  |
  Lung: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Lung |  |  |  |  | 1.1 [1.1 to 1.1] |

4. Secondary Outcome: Image Quality as Assessed by Tumour-To-Background Ratio Presented by Peptide Mass and Radioactivity Dose Ranges
Description: For each PET assessment image quality was quantitatively measured by the tumour-to-background ratio, obtained using the mean of all lesions tumour-to-backgrounds, for each of the following organs; liver, lymph nodes, bone and lungs. The tumour-to-background ratio was computed by SUVmean of the lesion divided by the SUVmean of the subject's reference tissue (tumour-free liver or aortic blood). A high tumour-to-background ratio indicates high effectiveness of 68Ga-satoreotide trizoxetan as a diagnostic agent. Tumour-to-background ratios are presented for primary site of GEP-NET and per organ by both peptide mass range and radioactivity dose range.
Time Frame: Day 1 and Days 16 to 22
Population: as for outcome 2
Measure: Median (Full Range); unit: Ratio
Arm/Group | Peptide Mass Dose Range 5-20 μg | Peptide Mass Dose Range 30-45 μg | Radioactivity Dose Range 40-80 MBq | Radioactivity Dose Range 100-140 MBq | Radioactivity Dose Range 160-200 MBq
Number analyzed (Participants) | 24 | 24 | 16 | 16 | 16
Ratio
  Primary Site: number analyzed (Participants) | 6 | 5 | 3 | 5 | 3
  Primary Site | 5.9 [2.28 to 45.84] | 7.1 [2.22 to 32.81] | 7.0 [2.22 to 45.84] | 7.1 [4.57 to 33.81] | 3.3 [2.28 to 32.81]
  Liver: number analyzed (Participants) | 18 | 18 | 13 | 10 | 13
  Liver | 4.1 [2.13 to 24.95] | 4.3 [3.05 to 29.33] | 4.3 [3.07 to 22.48] | 4.4 [3.10 to 24.95] | 4.1 [2.13 to 29.33]
  Lymph Nodes: number analyzed (Participants) | 14 | 14 | 8 | 9 | 11
  Lymph Nodes | 5.5 [2.55 to 16.98] | 5.2 [1.54 to 18.69] | 4.9 [3.50 to 18.69] | 5.3 [2.55 to 16.10] | 5.7 [1.54 to 13.70]
  Bone: number analyzed (Participants) | 1 | 1 | 0 | 1 | 1
  Bone | 12.7 [12.7 to 12.7] | 9.2 [9.2 to 9.2] |  | 12.7 [12.7 to 12.7] | 9.2 [9.2 to 9.2]
  Lung: number analyzed (Participants) | 1 | 0 | 0 | 0 | 1
  Lung | 1.1 [1.1 to 1.1] |  |  |  | 1.1 [1.1 to 1.1]

5. Secondary Outcome: Image Quality as Assessed by Independent Blinded Readers Quality Score
Description: A qualitative analysis of the image was assessed by 2 independent blinded readers using a quality score (performed as a back-up to the quantitative quality measured by tumour-to-background analysis). For each PET/CT and PET assessment, each reader performed a direct comparison of the 2 scans from Visit 2 and Visit 3. They noted which scan provided superior images based on overall image quality and lesion count and attributed a score for each assessment. The score for the assessment having superior images was set to "1", and score for the assessment not selected was set to "0". In case of equal quality, both assessments had a score of "1". The image quality score for PET/CT and PET readings as cumulative sum of readers' scores across all subjects by peptide mass and radioactivity dose range combination is presented. Score ranges from 0-16 with higher score indicating more assessments classed as superior.
Time Frame: Day 1 and Days 16 to 22
Population: Results are presented for the PP population which consisted of the first 24 randomised subjects who could be assessed and for whom no major protocol violations/deviations impacting primary endpoint results occurred. Only subjects with data available were included in the analysis. Note: image scores are presented as the cumulative sum of both readers' results across all subjects analysed per specified combination/visit; they do not represent summarised values.
Measure: Number; unit: Cumulative Sum of Readers' Scores
Arm/Group | Radioactivity Dose Range 40-80 MBq | Radioactivity Dose Range 100-140 MBq | Radioactivity Dose Range 160-200 MBq
Number analyzed (Participants) | 16 | 16 | 16
Cumulative Sum of Readers' Scores
  PET/CT: Peptide mass 5-20 μg (Visit 2): number analyzed (Participants) | 8 | 8 | 8
  PET/CT: Peptide mass 5-20 μg (Visit 2) | 9 | 10 | 10
  PET/CT: Peptide mass 30-45 μg (Visit 3): number analyzed (Participants) | 8 | 8 | 8
  PET/CT: Peptide mass 30-45 μg (Visit 3) | 13 | 14 | 13
  PET: Peptide mass 5-20 μg (Visit 2): number analyzed (Participants) | 8 | 8 | 8
  PET: Peptide mass 5-20 μg (Visit 2) | 7 | 14 | 13
  PET: Peptide mass 30-45 μg (Visit 3): number analyzed (Participants) | 8 | 8 | 8
  PET: Peptide mass 30-45 μg (Visit 3) | 11 | 15 | 13

6. Secondary Outcome: Lesion Maximum Standardised Uptake Value (SUVmax) Presented by Combination of Injected Peptide/Radioactivity Dose Ranges
Description: For each PET assessment, SUVmax was measured for each lesion, up to a maximum of 5 most avid lesions per organ that were confirmed by SoT assessment. In order to obtain a unique measure per organ, values of the SUVmax were computed within each of the following organs; liver, lymph nodes, bone and lungs. SUVmax results are presented for primary site of GEP-NET and per organ by each combination of injected peptide/radioactivity dose range.
Time Frame: Day 1 and Days 16 to 22
Population: as for outcome 2
Measure: Median (Full Range); unit: SUV
Arm/Group | Arm A: 5-20 μg/40-80 MBq | Arm A: 30-45 μg/100-140 MBq | Arm B: 5-20 μg/100-140 MBq | Arm B: 30-45 μg/160-200 MBq | Arm C: 5-20 μg/160-200 MBq | Arm C: 30-45 μg/40-80 MBq
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8
SUV
  Primary Site: number analyzed (Participants) | 2 | 2 | 3 | 2 | 1 | 1
  Primary Site | 90.3 [44.63 to 136.04] | 90.3 [43.34 to 137.34] | 24.5 [16.66 to 86.71] | 48.9 [11.93 to 85.78] | 14.2 [14.2 to 14.2] | 13.7 [13.7 to 13.7]
  Liver: number analyzed (Participants) | 5 | 5 | 5 | 5 | 8 | 8
  Liver | 24.2 [18.25 to 49.16] | 22.9 [18.01 to 59.83] | 9.5 [6.74 to 63.68] | 16.0 [9.56 to 78.43] | 12.4 [6.95 to 30.07] | 17.7 [10.62 to 30.28]
  Lymph Nodes: number analyzed (Participants) | 3 | 3 | 6 | 6 | 5 | 5
  Lymph Nodes | 24.7 [19.52 to 40.74] | 35.7 [16.69 to 41.11] | 28.5 [9.03 to 83.06] | 27.7 [5.25 to 53.79] | 13.8 [6.08 to 21.73] | 12.7 [6.15 to 21.33]
  Bone: number analyzed (Participants) | 0 | 0 | 1 | 1 | 0 | 0
  Bone |  |  | 57.5 [57.5 to 57.5] | 36.5 [36.5 to 36.5] |  |
  Lung: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Lung |  |  |  |  | 1.8 [1.8 to 1.8] |

7. Secondary Outcome: Lesion SUVmax Presented by Peptide Mass and Radioactivity Dose Ranges
Description: For each PET assessment, SUVmax was measured for each lesion, up to a maximum of 5 most avid lesions per organ that are confirmed by SoT assessment. In order to obtain a unique measure per organ, mean of the SUVmax was computed within each of the liver, lymph nodes, bone and lungs. SUVmax results are presented for primary site of GEP-NET and per organ by both peptide mass range and radioactivity dose range.
Time Frame: Day 1 and Days 16 to 22
Population: as for outcome 2
Measure: Median (Full Range); unit: SUV
Arm/Group | Peptide Mass Dose Range 5-20 μg | Peptide Mass Dose Range 30-45 μg | Radioactivity Dose Range 40-80 MBq | Radioactivity Dose Range 100-140 MBq | Radioactivity Dose Range 160-200 MBq
Number analyzed (Participants) | 24 | 24 | 16 | 16 | 16
SUV
  Primary Site: number analyzed (Participants) | 6 | 5 | 3 | 5 | 3
  Primary Site | 34.5 [14.19 to 136.04] | 43.3 [11.93 to 137.34] | 44.6 [13.67 to 136.04] | 43.3 [16.66 to 137.34] | 14.2 [11.93 to 85.78]
  Liver: number analyzed (Participants) | 18 | 18 | 13 | 10 | 13
  Liver | 15.6 [6.74 to 63.68] | 21.1 [9.56 to 78.43] | 20.0 [10.62 to 49.16] | 20.1 [6.74 to 63.68] | 13.3 [6.95 to 78.43]
  Lymph Nodes: number analyzed (Participants) | 14 | 14 | 8 | 9 | 11
  Lymph Nodes | 20.6 [6.08 to 83.06] | 20.3 [5.25 to 53.79] | 20.4 [6.15 to 40.74] | 32.6 [9.03 to 83.06] | 18.6 [5.25 to 53.79]
  Bone: number analyzed (Participants) | 1 | 1 | 0 | 1 | 1
  Bone | 57.5 [57.5 to 57.5] | 36.5 [36.5 to 36.5] |  | 57.5 [57.5 to 57.5] | 36.5 [36.5 to 36.5]
  Lung: number analyzed (Participants) | 1 | 0 | 0 | 0 | 1
  Lung | 1.8 [1.8 to 1.8] |  |  |  | 1.8 [1.8 to 1.8]

8. Secondary Outcome: Absolute Number of Lesions Detected by 68Ga-Satoreotide Trizoxetan Presented by Combination of Injected Peptide/Radioactivity Dose Range
Description: For each PET/CT and PET assessment, the absolute number of lesions detected by 68Ga-satoreotide trizoxetan were reported for each of the following anatomic sites; primary site of GEP-NET, liver, lymph nodes, axial/appendicular skeleton (bone) and lungs. The absolute number of lesions for PET/CT and PET readings for the 5 anatomic sites are presented by each combination of injected peptide/radioactivity dose range.
Time Frame: Day 1 and Days 16 to 22
Population: as for outcome 2
Measure: Median (Full Range); unit: Lesions
Arm/Group | Arm A: 5-20 μg/40-80 MBq | Arm A: 30-45 μg/100-140 MBq | Arm B: 5-20 μg/100-140 MBq | Arm B: 30-45 μg/160-200 MBq | Arm C: 5-20 μg/160-200 MBq | Arm C: 30-45 μg/40-80 MBq
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8
Lesions
  PET/CT: Primary Site | 1.0 [0 to 1] | 1.0 [0 to 1] | 0.0 [0 to 1] | 0.5 [0 to 1] | 1.0 [0 to 1] | 1.0 [0 to 1]
  PET/CT: Liver: number analyzed (Participants) | 8 | 8 | 7 | 7 | 8 | 8
  PET/CT: Liver | 8.5 [3 to 15] | 12.5 [3 to 22] | 8.0 [0 to 19] | 11.0 [0 to 21] | 14.5 [3 to 71] | 14.5 [3 to 93]
  PET/CT: Lymph Nodes: number analyzed (Participants) | 7 | 7 | 7 | 7 | 8 | 8
  PET/CT: Lymph Nodes | 4.0 [0 to 9] | 2.0 [0 to 6] | 4.0 [0 to 8] | 2.0 [0 to 12] | 6.0 [1 to 11] | 3.5 [1 to 10]
  PET/CT: Bone: number analyzed (Participants) | 3 | 3 | 7 | 7 | 4 | 4
  PET/CT: Bone | 2.0 [1 to 6] | 1.0 [1 to 5] | 1.0 [0 to 55] | 1.0 [1 to 43] | 2.0 [1 to 10] | 3.0 [2 to 6]
  PET/CT: Lung: number analyzed (Participants) | 4 | 4 | 5 | 5 | 3 | 3
  PET/CT: Lung | 0.0 [0 to 0] | 0.0 [0 to 0] | 0.0 [0 to 1] | 0.0 [0 to 2] | 0.0 [0 to 1] | 0.0 [0 to 0]
  PET: Primary Site | 1.0 [0 to 1] | 1.0 [0 to 1] | 1.0 [0 to 1] | 0.5 [0 to 1] | 1.0 [1 to 1] | 1.0 [1 to 1]
  PET: Liver: number analyzed (Participants) | 8 | 8 | 7 | 7 | 8 | 8
  PET: Liver | 7.5 [3 to 22] | 9.0 [3 to 23] | 8.0 [0 to 25] | 13.0 [0 to 26] | 14.0 [3 to 76] | 11.0 [3 to 78]
  PET: Lymph Nodes: number analyzed (Participants) | 7 | 7 | 7 | 7 | 8 | 8
  PET: Lymph Nodes | 4.0 [0 to 9] | 4.0 [0 to 10] | 3.0 [0 to 21] | 2.0 [0 to 18] | 6.5 [1 to 10] | 4.5 [1 to 8]
  PET: Bone: number analyzed (Participants) | 3 | 3 | 7 | 7 | 4 | 4
  PET: Bone | 1.0 [1 to 1] | 1.0 [0 to 1] | 1.0 [0 to 43] | 1.0 [0 to 46] | 3.5 [2 to 15] | 3.0 [1 to 13]
  PET: Lung: number analyzed (Participants) | 4 | 4 | 5 | 5 | 3 | 3
  PET: Lung | 0.5 [0 to 2] | 0.0 [0 to 1] | 0.0 [0 to 2] | 2.0 [0 to 4] | 2.0 [0 to 4] | 0.0 [0 to 0]

9. Secondary Outcome: Absolute Number of Lesions Detected by 68Ga-Satoreotide Trizoxetan Presented by Peptide Mass and Radioactivity Dose Ranges
Description: For each PET/CT and PET assessment, the absolute number of lesions detected by 68Ga-satoreotide trizoxetan were reported for each of the following anatomic sites; primary site of GEP-NET, lymph nodes, liver, axial/appendicular skeleton (bone) and lungs. The absolute number of lesions for PET/CT and PET readings for the 5 anatomic sites are presented by both peptide mass range and radioactivity dose range.
Time Frame: Day 1 and Days 16 to 22
Population: as for outcome 2
Measure: Median (Full Range); unit: Lesions
Arm/Group | Peptide Mass Dose Range 5-20 μg | Peptide Mass Dose Range 30-45 μg | Radioactivity Dose Range 40-80 MBq | Radioactivity Dose Range 100-140 MBq | Radioactivity Dose Range 160-200 MBq
Number analyzed (Participants) | 24 | 24 | 16 | 16 | 16
Lesions
  PET/CT: Primary Site | 1.0 [0 to 1] | 1.0 [0 to 1] | 1.0 [0 to 1] | 0.5 [0 to 1] | 1.0 [0 to 1]
  PET/CT: Liver: number analyzed (Participants) | 23 | 23 | 16 | 15 | 15
  PET/CT: Liver | 9.0 [0 to 71] | 13.0 [0 to 93] | 11.5 [3 to 93] | 11.0 [0 to 22] | 11.0 [0 to 71]
  PET/CT: Lymph Nodes: number analyzed (Participants) | 22 | 22 | 15 | 14 | 15
  PET/CT: Lymph Nodes | 4.5 [0 to 11] | 2.0 [0 to 12] | 4.0 [0 to 10] | 2.0 [0 to 8] | 4.0 [0 to 12]
  PET/CT: Bone: number analyzed (Participants) | 14 | 14 | 7 | 10 | 11
  PET/CT: Bone | 1.0 [0 to 55] | 1.5 [1 to 43] | 3.0 [1 to 6] | 1.0 [0 to 55] | 1.0 [1 to 43]
  PET/CT: Lung: number analyzed (Participants) | 12 | 12 | 7 | 9 | 8
  PET/CT: Lung | 0.0 [0 to 1] | 0.0 [0 to 2] | 0.0 [0 to 0] | 0.0 [0 to 1] | 0.0 [0 to 2]
  PET: Primary Site | 1.0 [0 to 1] | 1.0 [0 to 1] | 1.0 [0 to 1] | 1.0 [0 to 1] | 1.0 [0 to 1]
  PET: Liver: number analyzed (Participants) | 23 | 23 | 16 | 15 | 15
  PET: Liver | 9.0 [0 to 76] | 11.0 [0 to 78] | 10.0 [3 to 78] | 8.0 [0 to 25] | 13.0 [0 to 76]
  PET: Lymph Nodes: number analyzed (Participants) | 22 | 22 | 15 | 14 | 15
  PET: Lymph Nodes | 6.0 [0 to 21] | 4.0 [0 to 18] | 4.0 [0 to 9] | 3.5 [0 to 21] | 6.0 [0 to 18]
  PET: Bone: number analyzed (Participants) | 14 | 14 | 7 | 10 | 11
  PET: Bone | 1.5 [0 to 43] | 1.0 [0 to 46] | 1.0 [1 to 13] | 1.0 [0 to 43] | 2.0 [0 to 46]
  PET: Lung: number analyzed (Participants) | 12 | 12 | 7 | 9 | 8
  PET: Lung | 0.5 [0 to 4] | 0.0 [0 to 4] | 0.0 [0 to 2] | 0.0 [0 to 2] | 2.0 [0 to 4]

10. Secondary Outcome: Difference in Number of Lesions Detected by 68Ga-Satoreotide Trizoxetan Compared to Lesions Detected by SoT Presented by Combination of Injected Peptide/Radioactivity Dose Range
Description: For each PET/CT and PET assessment, the number of lesions detected by 68Ga-satoreotide trizoxetan and SoT (ceCT) were reported for each of the following anatomic sites; primary site of GEP-NET, lymph nodes, liver, axial/appendicular skeleton (bone) and lungs. The difference was calculated by number of lesions detected by 68Ga-satoreotide trizoxetan - number of lesions detected by ceCT scan. A positive difference indicates that more lesions were detected by 68Ga-satoreotide trizoxetan than by ceCT scan. A negative difference indicates that more lesions were detected by ceCT scan than by 68Ga-satoreotide trizoxetan. The difference in number of lesions for PET/CT and PET readings for the 5 anatomic sites are presented by each combination of injected peptide/radioactivity dose range.
Time Frame: Day 1 and Days 16 to 22
Population: as for outcome 2
Measure: Median (Full Range); unit: Lesions
Arm/Group | Arm A: 5-20 μg/40-80 MBq | Arm A: 30-45 μg/100-140 MBq | Arm B: 5-20 μg/100-140 MBq | Arm B: 30-45 μg/160-200 MBq | Arm C: 5-20 μg/160-200 MBq | Arm C: 30-45 μg/40-80 MBq
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8
Lesions
  PET/CT: Primary Site | 0.5 [-1 to 1] | 0.5 [-1 to 1] | 0.0 [-1 to 1] | 0.0 [0 to 1] | 0.5 [0 to 1] | 0.5 [0 to 1]
  PET/CT: Liver: number analyzed (Participants) | 8 | 8 | 7 | 7 | 8 | 8
  PET/CT: Liver | 6.0 [-3 to 13] | 9.0 [3 to 14] | 8.0 [-1 to 19] | 10.0 [0 to 21] | 4.0 [-3 to 53] | 5.5 [-5 to 75]
  PET/CT: Lymph Nodes: number analyzed (Participants) | 7 | 7 | 7 | 7 | 8 | 8
  PET/CT: Lymph Nodes | 2.0 [0 to 8] | 0.0 [-3 to 4] | 0.0 [-3 to 7] | 0.0 [-2 to 11] | 3.0 [1 to 11] | 1.0 [0 to 10]
  PET/CT: Bone: number analyzed (Participants) | 3 | 3 | 7 | 7 | 4 | 4
  PET/CT: Bone | 2.0 [1 to 6] | 1.0 [1 to 5] | 1.0 [0 to 43] | 1.0 [1 to 31] | 2.0 [1 to 10] | 3.0 [2 to 6]
  PET/CT: Lung: number analyzed (Participants) | 4 | 4 | 5 | 5 | 3 | 3
  PET/CT: Lung | 0.0 [0 to 0] | 0.0 [0 to 0] | 0.0 [-1 to 1] | 0.0 [-1 to 1] | 0.0 [0 to 1] | 0.0 [0 to 0]
  PET: Primary Site | 0.5 [-1 to 1] | 0.5 [-1 to 1] | 0.5 [0 to 1] | 0.0 [-1 to 1] | 1.0 [0 to 1] | 1.0 [0 to 1]
  PET: Liver: number analyzed (Participants) | 8 | 8 | 7 | 7 | 8 | 8
  PET: Liver | 4.0 [-3 to 22] | 5.5 [0 to 21] | 8.0 [-2 to 25] | 11.0 [0 to 26] | 5.0 [-3 to 58] | 5.0 [-8 to 60]
  PET: Lymph Nodes: number analyzed (Participants) | 7 | 7 | 7 | 7 | 8 | 8
  PET: Lymph Nodes | 2.0 [0 to 8] | 3.0 [0 to 10] | 1.0 [-2 to 18] | 1.0 [-2 to 13] | 5.5 [0 to 8] | 4.5 [-1 to 7]
  PET: Bone: number analyzed (Participants) | 3 | 3 | 7 | 7 | 4 | 4
  PET: Bone | 1.0 [1 to 1] | 1.0 [0 to 1] | 1.0 [0 to 31] | 1.0 [0 to 34] | 3.5 [2 to 15] | 3.0 [1 to 13]
  PET: Lung: number analyzed (Participants) | 4 | 4 | 5 | 5 | 3 | 3
  PET: Lung | 0.5 [0 to 2] | 0.0 [0 to 1] | 0.0 [-1 to 2] | 2.0 [-1 to 4] | 2.0 [0 to 4] | 0.0 [0 to 0]

11. Secondary Outcome: Difference in Number of Lesions Detected by 68Ga-Satoreotide Trizoxetan Compared to Lesions Detected by SoT Presented by Peptide Mass and Radioactivity Dose Ranges
Description: For each PET/CT and PET assessment, the number of lesions detected by 68Ga-satoreotide trizoxetan and SoT (ceCT) were reported for each of the following anatomic sites; primary site of GEP-NET, lymph nodes, liver, axial/appendicular skeleton (bone) and lungs. The difference was calculated by number of lesions detected by 68Ga-satoreotide trizoxetan - number of lesions detected by ceCT scan. A positive difference indicates that more lesions were detected by 68Ga-satoreotide trizoxetan than by ceCT scan. A negative difference indicates that more lesions were detected by ceCT scan than by 68Ga-satoreotide trizoxetan. The difference in number of lesions for PET/CT and PET readings for the 5 anatomic sites results are presented by both peptide mass range and radioactivity dose range.
Time Frame: Day 1 and Days 16 to 22
Population: as for outcome 2
Measure: Median (Full Range); unit: Lesions
Arm/Group | Peptide Mass Dose Range 5-20 μg | Peptide Mass Dose Range 30-45 μg | Radioactivity Dose Range 40-80 MBq | Radioactivity Dose Range 100-140 MBq | Radioactivity Dose Range 160-200 MBq
Number analyzed (Participants) | 24 | 24 | 16 | 16 | 16
Lesions
  PET/CT: Primary Site | 0.0 [-1 to 1] | 0.0 [-1 to 1] | 0.5 [-1 to 1] | 0.0 [-1 to 1] | 0.0 [0 to 1]
  PET/CT: Liver: number analyzed (Participants) | 23 | 23 | 16 | 15 | 15
  PET/CT: Liver | 7.0 [-3 to 53] | 10.0 [-5 to 75] | 5.5 [-5 to 75] | 8.0 [-1 to 19] | 10.0 [-3 to 53]
  PET/CT: Lymph Nodes: number analyzed (Participants) | 22 | 22 | 15 | 14 | 15
  PET/CT: Lymph Nodes | 2.0 [-3 to 11] | 1.0 [-3 to 11] | 2.0 [0 to 10] | 0.0 [-3 to 7] | 1.0 [-2 to 11]
  PET/CT: Bone: number analyzed (Participants) | 14 | 14 | 7 | 10 | 11
  PET/CT: Bone | 1.0 [0 to 43] | 1.5 [1 to 31] | 3.0 [1 to 6] | 1.0 [0 to 43] | 1.0 [1 to 31]
  PET/CT: Lung: number analyzed (Participants) | 12 | 12 | 7 | 9 | 8
  PET/CT: Lung | 0.0 [-1 to 1] | 0.0 [-1 to 1] | 0.0 [0 to 0] | 0.0 [-1 to 1] | 0.0 [-1 to 1]
  PET: Primary Site | 1.0 [-1 to 1] | 1.0 [-1 to 1] | 1.0 [-1 to 1] | 0.5 [-1 to 1] | 1.0 [-1 to 1]
  PET: Liver: number analyzed (Participants) | 23 | 23 | 16 | 15 | 15
  PET: Liver | 6.0 [-3 to 58] | 6.0 [-8 to 60] | 4.5 [-8 to 60] | 6.0 [-2 to 25] | 8.0 [-3 to 58]
  PET: Lymph Nodes: number analyzed (Participants) | 22 | 22 | 15 | 14 | 15
  PET: Lymph Nodes | 4.5 [-2 to 18] | 3.5 [-2 to 13] | 4.0 [-1 to 8] | 2.0 [-2 to 18] | 5.0 [-2 to 13]
  PET: Bone: number analyzed (Participants) | 14 | 14 | 7 | 10 | 11
  PET: Bone | 1.5 [0 to 31] | 1.0 [0 to 34] | 1.0 [1 to 13] | 1.0 [0 to 31] | 2.0 [0 to 34]
  PET: Lung: number analyzed (Participants) | 12 | 12 | 7 | 9 | 8
  PET: Lung | 0.0 [-1 to 4] | 0.0 [-1 to 4] | 0.0 [0 to 2] | 0.0 [-1 to 2] | 2.0 [-1 to 4]

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events (AEs) were recorded from Day 1 up to 14 days after the last dose of investigational imaging product (up to 36 days overall).
Description: All subjects included in the Safety Population analysis received 2 injections of 68Ga-satoreotide trizoxetan during the study. AEs were allocated to each combination of injected peptide/radioactivity dose range according to the following rule: AEs were allocated to the last dose of 68Ga-satoreotide trizoxetan received, based on AE start date/time.
Groups:
- Overall: Total number of AEs experienced across all Arms.
Arm/Group | Arm A: 5-20 μg/40-80 MBq | Arm A: 30-45 μg/100-140 MBq | Arm B: 5-20 μg/100-140 MBq | Arm B: 30-45 μg/160-200 MBq | Arm C: 5-20 μg/160-200 MBq | Arm C: 30-45 μg/40-80 MBq | Overall
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/9 | 0/9 | 0/10 | 0/10 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/9 | 0/9 | 0/10 | 0/10 | 0/27
Other Adverse Events (participants affected / at risk) | 2/8 | 4/8 | 4/9 | 6/9 | 3/10 | 5/10 | 18/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: 5-20 μg/40-80 MBq (N=8) | Arm A: 30-45 μg/100-140 MBq (N=8) | Arm B: 5-20 μg/100-140 MBq (N=9) | Arm B: 30-45 μg/160-200 MBq (N=9) | Arm C: 5-20 μg/160-200 MBq (N=10) | Arm C: 30-45 μg/40-80 MBq (N=10) | Overall (N=27)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Administration site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (3)
Feeling cold (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (3)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 5 (6)
Blood potassium increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood urine present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Basedow's disease (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
In each injected peptide/radioactivity dose combination for outcome measures 1, 3 and 6, the number of subjects with lesions in the primary site of GEP-NET, bone and lung was too small (0 to 3) to allow for a meaningful interpretation of the results. Similarly, in each category of peptide mass range and radioactivity dose range for outcome measures 2, 4 and 7, the number of subjects with lesions in bone and lung was too small (0 to 2) to allow for a meaningful interpretation of the results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-05-20): https://cdn.clinicaltrials.gov/large-docs/17/NCT03220217/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-28): https://cdn.clinicaltrials.gov/large-docs/17/NCT03220217/SAP_001.pdf